CLINICAL TRIAL: NCT07299825
Title: Phase 2 Study of A166 in HER2-positive Metastatic Breast Cancer Patients Who Were Previously Treated With TOP1-ADCs
Brief Title: A Study of A166 in Patients With HER2-Positive Unresectable or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL166-II-08
Record Dates: First submitted 2025-12-03; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Her 2 Positive Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A166 (Experimental): A166 is administered intravenously at a dose of 4.8 mg/kg every 21 (±3) days (q3w).
  Interventions: Drug: A166

INTERVENTIONS:
Drug: A166 — intravenous(IV) infusion (Q3W)

SUMMARY:
Evaluation of the efficacy of A166 in Patients with HER2-Positive unresectable or metastatic breast cancer previously treated with TOP1 inhibitor Antibody-Drug Conjugates

DETAILED DESCRIPTION:
This study will evaluate the efficacy of A166 in patients with HER2-positive unresectable or metastatic breast cancer previously treated with TOP1 inhibitor Antibody-Drug Conjugates.

A166 will be administered every 3 weeks (Q3W) intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years and ≤ 75 years when signing the informed consent form.
2. Breast cancer patients by histopathology and/or cytology documented.
3. In the advanced or metastatic stage, having received no more than 5 lines of systemic therapy, one of which must include a HER2 ADC with a topoisomerase inhibitor payload.
4. Patients must have experienced disease progression or intolerance during or after the most recent treatment prior to randomization.
5. At least one measurable lesion according to RECIST 1.1 criteria.

Exclusion Criteria:

1. Previous treatment with A166 or any HER2-targeted antibody-drug conjugate (ADC) with a microtubule inhibitor payload.
2. Known history of severe hypersensitivity to other monoclonal antibodies, or allergy to A166 or their components.
3. Permanent discontinuation of trastuzumab or its biosimilars due to any toxicity in prior treatments.
4. Presence of severe corneal epithelial disease at baseline; or inability to perform daily activities without contact lenses.
5. Presence of spinal cord compression or clinically active central nervous system (CNS) metastases.
6. Other conditions considered by the investigator to make the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Within 24 months of last patient enrolled
  ORR is defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed by investigator per RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Within 24 months of last patient enrolled
  PFS, 6-month PFS, 12-month PFS.PFS as assessed by investigator according to RECIST v 1.1
Overall survival (OS) | Within 48 months of last patient enrolled
  OS, 1-year survival rate, 1.5-year survival rate, and 2-year survival rate.OS defined as time from inclusion until death
Disease control rate(DCR) | Within 24 months of last patient enrolled
  DCR is defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by investigator per RECIST 1.1
Duration of response(DOR) | Within 24 months of last patient enrolled
  DoR is defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by investigator or death due to any cause, whichever occurs first.
Clinical Benefit Rate (CBR) | Within 24 months of last patient enrolled
  CBR is defined as a patient having a best overall response of a complete response (CR), partial response (PR), or stable disease for at least 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial Cancer Hospital, Zhenzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No